CLINICAL TRIAL: NCT00727831
Title: Phase I Trial of Escalating High Dose Methotrexate Supported by Glucarpidase to Treat Patients With Primary Central Nervous Lymphoma (PCNSL)
Brief Title: Methotrexate, Glucarpidase, and Leucovorin in Treating Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000599206; CRUK-BRD/07/004; 2007-002570-58; EU-20861
Record Dates: First submitted 2008-08-01; First posted 2008-08-04 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Chemotherapeutic Agent Toxicity; Lymphoma; Mucositis; Neurotoxicity
Keywords: neurotoxicity; chemotherapeutic agent toxicity; mucositis; primary central nervous system non-Hodgkin lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Mucositis; Neurotoxicity Syndromes; Lymphoma, Large B-Cell, Diffuse | interventions — glucarpidase; Leucovorin; Methotrexate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: glucarpidase
Drug: leucovorin calcium
Drug: methotrexate
Other: laboratory biomarker analysis
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate and leucovorin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Glucarpidase may help return the level of methotrexate in the blood to a safe range. Giving high-dose methotrexate together with glucarpidase and leucovorin may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of methotrexate when given together with glucarpidase and leucovorin in treating patients with newly diagnosed primary central nervous system lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the dose-limiting toxicity of methotrexate (MTX) when given in combination with glucarpidase in patients with newly diagnosed primary CNS lymphoma (PCNSL).
* To determine the incidence of immediate reactions related to the use of glucarpidase in these patients.
* To define a safer, more practical, and simpler regimen for delivering multiple courses of high-dose MTX using glucarpidase and 'short' leucovorin calcium rescue in these patients.
* To monitor quality of life and mental function during and after therapy in these patients.

Secondary

* To use this regimen as a platform for phase III studies in PCNSL.
* To record disease response, duration of response, and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of high-dose methotrexate (HD-MTX).

Patients receive HD-MTX IV over 4 hours on day 1. Beginning 22 hours after the start of HD-MTX, patients receive glucarpidase IV over 15 minutes on day 2 followed by leucovorin calcium orally or IV on days 2-7. Treatment repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Within 2-4 weeks after completion of study treatment, patients achieving maximum response are stratified according to age (< 60 years vs ≥ 60 years) and may undergo whole brain radiotherapy (WBRT) once daily, 5 days a week, for 3 to 5 weeks.

Patients undergo blood sample collection periodically to assess glucarpidase antibodies and MTX levels.

Patients are assessed for mucositis incidence and severity periodically, and complete quality of life assessments using the EORTC QLQ-30 questionnaire and the Mini-Mental State questionnaire at baseline, during, and after completion of study.

After completion of study treatment, patients are followed at 6 weeks after WBRT, every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed primary CNS lymphoma (PCNSL)

  * Previously untreated disease
  * Diffuse large B-cell lymphoma histology
* Must be clinically eligible to receive standard 3 g/m² methotrexate if outside trial
* No clinically significant effusions or edema

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-3
* Neutrophils ≥ 1 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin < 1.5 times upper limit of normal
* Glomerular filtration rate (initially measured by EDTA/isotope method) ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy

Exclusion criteria:

* HIV positivity
* Dementia or neurological dysfunction not considered to be due to the PCNSL
* Other serious or uncontrolled medical conditions
* Prior malignancy, except adequately treated nonmelanoma skin cancer or carcinoma in situ

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic chemotherapy
* No concurrent prophylactic antibiotics
* No concurrent co-trimoxazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Immediate toxicity (incidence of reactions to glucarpidase) as determined by the NCI CTC
Incidence and severity of renal dysfunction as determined by the NCI CTC
Incidence and severity of mucositis as determined by the NCI CTC and WHO mucositis grading scale
Incidence and severity of CNS toxicity and neurocognitive changes taken from patients' medical records and measured using the Mini-Mental State questionnaire and MRI data

SECONDARY OUTCOMES:
Hematological toxicity (i.e., number of courses of therapy associated with neutrophils < 0.5 x 10e9/L or platelets < 50 x 10e9/L as measured by routine blood counts)
Incidence of infection (i.e., number of days with fever ≥ 38 C° measured by clinical examination and days of intravenous antibiotics taken from patients' medical records)
Number of inpatient days taken from patients' medical records
Disease response and remission rates measured by serial MRI scanning (and eye examination and lumbar puncture if necessary)
Disease outcome, time to progression, and overall survival at 2 years from start of therapy measured by clinical examination and serial MRI scanning
Relative dose intensity
Methotrexate levels post-glucarpidase (expressed as a clinically important reduction, which is defined as a methotrexate level of < 1 μmol/L in all post-glucarpidase samples)
Incidence of antibodies to glucarpidase measured serologically at the start of each methotrexate course and at follow-up visits if present during therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roderick Johnson, MD, Principal Investigator — Leeds General Infirmary
Locations (2):
- United Kingdom (2):
  - Leeds General Infirmary, Leeds, England
  - Torbay Hospital, Torquay, England